CLINICAL TRIAL: NCT00712088
Title: Project ICARE: Intervening for Community Awareness, Respect, & Empowerment - Behavioral Intervention to Reduce Sexual Risk Behavior of African American Men Who Have Sex With Men
Brief Title: Project ICARE: Intervening for Community Awareness, Respect, & Empowerment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Howard Brown Health Center (Other); University of Illinois at Chicago (Other); South Side Help Center (Unknown); Chicago Department of Public Health (Other Government)
Responsible Party: David McKirnan, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-5159
Record Dates: First submitted 2008-06-03; First posted 2008-07-09 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections
Keywords: HIV; Unsafe Sex; High Risk Sex; HIV Prevention; African-American; gay; bisexual; intervention trial
MeSH Terms: conditions — HIV Infections; Unsafe Sex; Homosexuality; Bisexuality

ARMS (2):
- 1: Group Intervention (Experimental): Group level intervention
  Interventions: Behavioral: Project ICARE
- 2: HCT (Active Comparator): Offer of HIV counseling and testing
  Interventions: Behavioral: HCT

INTERVENTIONS:
Behavioral: Project ICARE — Group-level intervention (Project ICARE)
  Other Names: Intervening for Community Awareness, Respect, & Empowerment
  Arms: 1: Group Intervention
Behavioral: HCT — Offer of HIV counseling and testing
  Arms: 2: HCT

SUMMARY:
This project will test the efficacy of a behavioral intervention to reduce sexual risk for HIV infection among African American Men who Have Sex with Men (MSM).

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older;
* Self-identify as African American
* Understand and read English;
* Live within the Chicago area;
* Report at least two (male or female) sex partners in the past three months, and unprotected anal sex with at least one male sex partner in the past three months.

Exclusion Criteria:

* Have been diagnosed with HIV within the past three months (to allow for psychological and behavioral adjustment following an initial HIV diagnosis);
* Have a specific plan to move from the Chicago area within the next nine months;
* Report active injection drug use other than hormones or steroids.
* Participated in the intervention video or the pilot phase of this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Unprotected Sex | past three months

CONTACTS AND LOCATIONS:
Overall Officials: David McKirnan, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Howard Brown Health Center, Chicago, Illinois, United States